CLINICAL TRIAL: NCT02732288
Title: Exploratory Study of Melatonin Induced Sleep Regularization in Severe Brain Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interrupted by Covid-19
Sponsor: Rockefeller University (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NSC-0894
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Disorders of Consciousness
MeSH Terms: conditions — Consciousness Disorders | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin, brain injured patients (Experimental): Melatonin 3mg, orally, at 8pm, daily for 3 months
  Interventions: Dietary Supplement: melatonin
- Healthy volunteers (Experimental): Melatonin 3mg, orally, at 8pm
  Interventions: Dietary Supplement: melatonin

INTERVENTIONS:
Dietary Supplement: melatonin — After measuring the subject's own timing of release of melatonin, subjects will be provided a dose of melatonin at 8pm to test the effects on the electrical activity of sleep, measured using electroencephalography. The same intervention will be given to healthy, non-brain injured controls.

SUMMARY:
Patients with severe brain injuries often have slow accumulating recoveries of function. In ongoing studies, we have discovered that elements of electrical activity during sleep may correlate with the level of behavioral recovery observed in patients. It is unknown whether such changes are causally linked to behavioral recovery. Sleep processes are, however, associated with several critical processes supporting the cellular integrity of neurons and neuronal mechanisms associated with learning and synaptic modifications. These known associations suggest the possibility that targeting the normalization of brain electrical activity during sleep may aid the recovery process. A well-studied mechanism organizing the pattern of electrical activity that characterizes sleep is the body's release of the substance melatonin. Melatonin is produced in the brain and released at a precise time during the day (normally around 8-10PM) to signal the brain to initiate aspects of the sleep process each day. Ongoing research by other scientists has demonstrated that providing a small dose of melatonin can improve the regular pattern of sleep and help aid sleep induction. Melatonin use has been shown to be effective in the treatment of time change effects on sleep ("jet lag") and mood disturbances associated with changes in daily light cues such as seasonal affective disorder. We propose to study the effects of melatonin administration in patients with severe structural brain injuries and disorders of consciousness. We will measure the patient's own timing of release of melatonin and provide a dose of melatonin at night to test the effects on the electrical activity of sleep over a three month period. In addition to brain electrical activity we will record sleep behavioral data and physical activity using activity monitors worn by the patients. Patient subjects in this study will be studied twice during the three month period in three day inpatient visits where they will undergo video monitoring and sampling of brain electrical activity using pasted electrodes ("EEG"), hourly saliva sampling for one day, and participation in behavioral testing.

DETAILED DESCRIPTION:
Patients with severe brain injuries often have slow accumulating recoveries of function. Recently, the National Institute for Disability and Rehabilitation Research (NIDRR) published data on their long-term outcomes of over 9,000 patients, 400 of which suffered disorders of consciousness (Nakase-Richardson et al. 2012). Patients were followed for 1, 2, and 5 year outcomes and several important and unexpected results were obtained: a large majority of patients initially in minimally conscious state (MCS) continued to improve recovering consciousness within a year and recovery was demonstrated to continue at the 2 and 5 year timepoints for as many as 20% of patients. In these cases outcomes included vocational reentry. Other studies have confirmed that MCS recovery can occur over long-time periods and lead to good outcomes or significant recovery of meaningful cognitive function despite enduring convalesce in MCS (Luaute et al. 2010, Lammi et al. 2005).

In ongoing studies we have discovered that elements of electrical activity during sleep may correlate with the level of behavioral recovery observed in patients (Forgacs et al. 2014, Thengone et al. 2012). It is unknown, however, whether such changes are causally linked to behavioral recovery. Forgacs et al. 2014 showed a cross- sectional relationship between retention of key elements of sleep EEG architecture and behavioral level. Thengone et al. 2012 correlated longitudinal changes in sleep architecture and quantitative spectral measures with behavioral recovery in 4 patients with severe brain injuries. No studies, however, have used an instrumental causal design to address whether improvement in sleep architecture can be promoted in patients with severe brain injuries and if so, whether or not changes in wakeful behavioral level are causally linked to such instrumentally generated changes in sleep.

Sleep processes are associated with several critical processes supporting the cellular integrity of neurons and neuronal mechanisms associated with learning and synaptic modifications giving face validity to this approach. (Steriade, 1999; Tononi and Cirelli, 2012). For example, studies in healthy volunteers (Huber et al. 2004) have provided evidence that local spindle density changes are associated with learning of specific information over sleep periods and can be topographically related to cortical populations engaged by the wakeful learning process. Additional evidence indicates that recovery of spindles within the electrical architecture of sleep is more associated with recovery of motor function in stroke (Gottselig, 2002). Collectively, although only a limited number of studies exist there is a biological basis for improvement in sleep architecture to potentially drive recovery and reorganization of brain networks organizing wakeful behavior.

These known associations suggest the possibility that targeting the normalization of brain electrical activity during sleep may aid the recovery process. In fact, in one human subject studied here in our program, central thalamic deep brain stimulation (CT-DBS) applied beginning 20 years after severe traumatic brain injury (TBI) correlated with a normalization of sleep architecture beginning at the time after exposure to continuous DBS. These findings strongly suggest a link between increased driving of synaptic activity during the day and modification of sleep processes as this subject was only exposed to CT-DBS during daytime hours (Adams et al 2014). These findings improve the likelihood that there is a bi-directional causal relationship sleep dynamics and wakeful brain dynamics as linked to changes in behavior. Thus, the working hypothesis of the present study is that causal intervention to normalize sleep processes in patients with severe brain injuries may aid recovery of behavioral function.

A well-studied mechanism organizing the normal patterns of electrical activity that characterizes sleep is the body's release of the substance melatonin. Melatonin is produced in the brain and released at a precise time during the day (normally around 8-10PM) to signal the brain to initiate aspects of the sleep process each day (Dijk, 1997). It is possible to exogenously trigger and drive melatonin signaling of sleep processes and initiation of sleep via oral dosing of the agent (Lewy et al. 1992). Use of oral melatonin supplements is common for pre- treatment of expected travel delay sleep disturbances ("jet lag") and has been investigated in treatment of mood disorders (Lewy et al. 1996).

Thus, we propose to study the effects of melatonin administration in patients with severe structural brain injuries and disorders of consciousness. An existing, though small, literature supports the probable success of this study; in neurodegenerative patients melatonin supplementation has shown modest benefit in improving some cognitive and noncognitive symptoms (Riemersma-van der Lek et al. 2008). Pediatric patients with traumatic brain injuries have been considered for treatment with melatonin based on similar considerations (Keegan et al. 2013)

What will we do: We will measure the patient's own timing of release of melatonin and provide a dose of melatonin at a standard time at night (8PM) to test the effects on the electrical activity of sleep over a three month period. In addition to brain electrical activity, we will record sleep behavioral data and physical activity using activity monitors worn by the patients. Patient subjects in this study will be studied twice during the three month period in three day inpatient visits where they will undergo video monitoring and sampling of brain electrical activity using pasted electrodes ("EEG"), hourly saliva sampling for one day, and participate in behavioral testing.

Why are the risks proportionate? Melatonin is very safe and has a limited and known adverse effect profile (Buscemi at al. 2004) Melatonin does not accumulate and can be stopped. We will carefully monitor the first dose during an in-patient stay. Moreover, from an ethical frame there is in this study a clear intention to treat. If our hypothesis is supported patients will meaningfully improve in function.

ELIGIBILITY:
Inclusion Criteria for subjects:

* Subject's legally authorized representative must be fluent in English
* Subject must have been able to speak English prior to the brain injury occurrence
* Subject must have previously participated in the NSC-0764 study at Rockefeller University Hospital or New York Presbyterian-Cornell
* Subject must be diagnosed with a severe nonprogressive brain injury
* Subject must be medically stable
* Subject must be between 18 and 65 years of age
* Male and female subjects accepted
* Subject must have previously participated in studies with EEG data that identify elements of sleep architecture (evidence of components of at least 1 of the following: Stage 2 features (e.g. spindles K complexes, or vertex waves) or stage 3 features (e.g. slow waves), including the NSC-0764 study, and this data must be available to the PI.

HEALTHY VOLUNTEERS: case matched to the study population +/- 5 years; fluent in English; ability to sit still for several consecutive hours; must sleep normal hours consistently (approximately 10 pm - about 6 am) and not be a shift worker

Exclusion Criteria for subjects:

* Refractory generalized seizures
* Ventilator dependency
* Evidence of Alzheimer's Disease or dementia preinjury
* Currently taking melatonin
* Dialysis dependency
* Premorbid neuropsychiatric history (Axis I requiring prior hospitalization)
* History of severe asthma (requiring hospitalization)
* Participation in any investigational trial within 30 days prior to enrollment in this study
* History of any sleep disorder or restless leg syndrome pre-injury
* Medical history, physical examination, or laboratory findings suggestive of any other medical or psychological condition that would, in the opinion of the principal investigator, make the candidate ineligible for the study

HEALTHY VOLUNTEERS: current or past medical history of any neurological disease or cardiovascular disease, sleep disorder, teeth grinding or restless leg syndrome (RLS); taking any medications with any neurologic effects, any medical condition that disrupts sleep; participation in NSC-0764; Body Mass Index (BMI) > 30 kg/m2;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-05; Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Changes in in sleep/wake architecture following melatonin administration as assessed by time domain analysis of sleep EEG | baseline, 3 months

SECONDARY OUTCOMES:
quantitative measures of EEG spectral content | baseline, 3 months
Changes in wakeful behavior level | baseline, 3 months
  Scales include: Coma Recovery Scale (CRS) and Confusion Assessment Protocol (CAP)
Activity levels captured by Actigraph device | baseline, 3 months
  Actigraph is a wearable motion detector used to monitor and track activity and sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Schiff, MD, Principal Investigator — Weill Cornell Medical College/ Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luaute J, Maucort-Boulch D, Tell L, Quelard F, Sarraf T, Iwaz J, Boisson D, Fischer C. Long-term outcomes of chronic minimally conscious and vegetative states. Neurology. 2010 Jul 20;75(3):246-52. doi: 10.1212/WNL.0b013e3181e8e8df. Epub 2010 Jun 16. PMID 20554940
- [Background] Lammi MH, Smith VH, Tate RL, Taylor CM. The minimally conscious state and recovery potential: a follow-up study 2 to 5 years after traumatic brain injury. Arch Phys Med Rehabil. 2005 Apr;86(4):746-54. doi: 10.1016/j.apmr.2004.11.004. PMID 15827927
- [Background] Forgacs PB, Conte MM, Fridman EA, Voss HU, Victor JD, Schiff ND. Preservation of electroencephalographic organization in patients with impaired consciousness and imaging-based evidence of command-following. Ann Neurol. 2014 Dec;76(6):869-79. doi: 10.1002/ana.24283. Epub 2014 Oct 24. PMID 25270034
- [Background] Steriade M. Coherent oscillations and short-term plasticity in corticothalamic networks. Trends Neurosci. 1999 Aug;22(8):337-45. doi: 10.1016/s0166-2236(99)01407-1. PMID 10407416
- [Background] Tononi G, Cirelli C. Time to be SHY? Some comments on sleep and synaptic homeostasis. Neural Plast. 2012;2012:415250. doi: 10.1155/2012/415250. Epub 2012 Apr 29. PMID 22619736
- [Background] Huber R, Ghilardi MF, Massimini M, Tononi G. Local sleep and learning. Nature. 2004 Jul 1;430(6995):78-81. doi: 10.1038/nature02663. Epub 2004 Jun 6. PMID 15184907
- [Background] Nakase-Richardson R, Whyte J, Giacino JT, Pavawalla S, Barnett SD, Yablon SA, Sherer M, Kalmar K, Hammond FM, Greenwald B, Horn LJ, Seel R, McCarthy M, Tran J, Walker WC. Longitudinal outcome of patients with disordered consciousness in the NIDRR TBI Model Systems Programs. J Neurotrauma. 2012 Jan 1;29(1):59-65. doi: 10.1089/neu.2011.1829. Epub 2011 Aug 4. PMID 21663544
- [Background] Gottselig JM, Bassetti CL, Achermann P. Power and coherence of sleep spindle frequency activity following hemispheric stroke. Brain. 2002 Feb;125(Pt 2):373-83. doi: 10.1093/brain/awf021. PMID 11844737
- [Background] Dijk DJ, Cajochen C. Melatonin and the circadian regulation of sleep initiation, consolidation, structure, and the sleep EEG. J Biol Rhythms. 1997 Dec;12(6):627-35. doi: 10.1177/074873049701200618. PMID 9406038
- [Background] Lewy AJ, Ahmed S, Jackson JM, Sack RL. Melatonin shifts human circadian rhythms according to a phase-response curve. Chronobiol Int. 1992 Oct;9(5):380-92. doi: 10.3109/07420529209064550. PMID 1394610
- [Background] Lewy AJ, Ahmed S, Sack RL. Phase shifting the human circadian clock using melatonin. Behav Brain Res. 1996;73(1-2):131-4. doi: 10.1016/0166-4328(96)00084-8. PMID 8788490
- [Background] Riemersma-van der Lek RF, Swaab DF, Twisk J, Hol EM, Hoogendijk WJ, Van Someren EJ. Effect of bright light and melatonin on cognitive and noncognitive function in elderly residents of group care facilities: a randomized controlled trial. JAMA. 2008 Jun 11;299(22):2642-55. doi: 10.1001/jama.299.22.2642. PMID 18544724
- [Background] Keegan LJ, Reed-Berendt R, Neilly E, Morrall MC, Murdoch-Eaton D. Effectiveness of melatonin for sleep impairment post paediatric acquired brain injury: evidence from a systematic review. Dev Neurorehabil. 2014 Oct;17(5):355-62. doi: 10.3109/17518423.2012.741147. Epub 2013 Oct 8. PMID 24102301
- [Background] Buscemi N, Vandermeer B, Pandya R, Hooton N, Tjosvold L, Hartling L, Baker G, Vohra S, Klassen T. Melatonin for treatment of sleep disorders. Evid Rep Technol Assess (Summ). 2004 Nov;(108):1-7. doi: 10.1037/e439412005-001. No abstract available. PMID 15635761